CLINICAL TRIAL: NCT01313832
Title: The Effect of Remote Ischemic Preconditioning on the Ischemic Reperfusion Injury in Infants With Ventricular Septal Defect and Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H-1012-120-345
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Ventricular Septal Defect; Pulmonary Hypertension
Keywords: ventricular septal defect; remote ischemic preconditioning; pulmonary hypertension; infant with ventricular septal defect and pulmonary hypertension
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- remote ischemic preconditioning (Experimental)
  Interventions: Other: remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Other: remote ischemic preconditioning (RIPC) — RIPC will be performed by 5-min cycles of lower limb ischemia reperfusion using blood pressure cuff

SUMMARY:
Intraoperative myocardial and pulmonary protection is important for better outcome after cardiac surgery. Ischemic preconditioning is one of organ protective strategies against ischemia-reperfusion injury by applying brief ischemia to the target organ before a subsequent critical ischemia, and its effect has been confirmed. However, its clinical application is not easy because ischemic insult may aggravate the function of vulnerable organ.

On the other hand, remote ischemic preconditioning (RIPC) is another protective approach by applying ischemia to other less vulnerable organ such as skeletal muscle before critical ischemia-reperfusion injury to heart. The effect of RIPC has been well demonstrated in adults and children. However, Little is known about the effect of remote ischemic precondition on the pediatric myocardium to ischemia and reperfusion injury. The effect of RIPC on the children remains to be further evaluated because the degree of ischemia-reperfusion injury is different according to age, cardiac pathology and cyanosis. In addition, the previous report on children dealt with a diverse range of congenital heart defects with a wide age range. The purpose of this study was to evaluate the effect of RIPC on myocardial and pulmonary protection in infants with pulmonary hypertension who need repair of simple ventricular septal defect.

ELIGIBILITY:
Inclusion Criteria:

* perimembranous or muscular outlet or muscular inlet ventricular septal defect
* pulmonary hypertension (+)
* infant (<1 year)

Exclusion Criteria:

* subarterial ventricular defect
* chromosomal defect
* airway or parenchymal lung disease
* blood disorder
* anticipation of cardiac muscle resection

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
troponin level | within the 1 day after operation
  troponin level will be checked 1, 6, 12 and 24 hours after operation. After making a graph for troponin-time, area under curve will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Park YH, Byon HJ, Kim HS, Kim CS, Kim JT. Effect of remote ischaemic preconditioning on ischaemic-reperfusion injury in pulmonary hypertensive infants receiving ventricular septal defect repair. Br J Anaesth. 2012 Feb;108(2):223-8. doi: 10.1093/bja/aer388. Epub 2011 Dec 8. PMID 22157844